CLINICAL TRIAL: NCT06861660
Title: Digitally Prompted Parenting: A Text Message Parent-Based Alcohol Intervention for Incoming College Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Responsible Party: Principal Investigator, Dr. Joseph LaBrie, Principal Investigator, Loyola Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R34AA031358-01A1 (NIH)
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study conditions are randomly assigned and the intervention delivery is automated. Senior members of the research team will have a record of the participants randomized to each condition, but the delivery of intervention content is automated. Junior members of the research team responsible for sending follow-up survey reminders will not be aware of participant condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitally Prompted Parenting (Experimental): Parents of participating first-year college students in this intervention arm will receive a series of prewritten text messages during the first 10 weeks of college. Parents can personalize these messages before sending them directly to their student, who is the study participant, with the goal of reducing alcohol-related risks.
  Interventions: Behavioral: Digitally Prompted Parenting
- Active Control (Active Comparator): Parents of participating first-year college students in this arm of the study will receive access to the Parent Handbook during the summer before matriculation and three booster emails that summarize its key points after matriculation.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Digitally Prompted Parenting — Parents will receive an email invitation to sign up for Digitally Prompted Parenting, a text message-delivered PBI. Parents set up an account and input information about themselves and their student, which will customize the text messages they receive. Parents will receive at least two text prompts per week for the first 10 weeks of their student's first semester in college. These texts will (1) prompt parents to call their student to discuss the past week and week ahead, and (2) prompt parents to send an alcohol-specific risk reducing text to their student.
  Arms: Digitally Prompted Parenting
Behavioral: Active Control — Parents will receive an email that explains the Parent Handbook intervention and includes a link to a website where the Handbook is embedded. They will also receive three booster emails summarizing the key points of the intervention. Parents can review both the Parent Handbook and the booster emails at their own pace.
  Arms: Active Control

SUMMARY:
This pilot randomized controlled trial (RCT) will evaluate both the feasibility and efficacy of Digitally Prompted Parenting (DPP), a text-message based parent intervention (tm-PBI) designed to prevent and reduce alcohol use among first-year college students. In this study, parents of incoming first-year students will receive risk-reducing text messages during the first 10 weeks of the Fall semester, which they can forward to their students. The trial uses a longitudinal design to compare drinking outcomes between students whose parents receive the DPP messages and those whose parents receive an established alcohol PBI (the active control condition). The investigators hypothesize that students in the DPP group will report lower levels of alcohol use and fewer alcohol-related consequences after the intervention compared to those in the active control group.

ELIGIBILITY:
Inclusion Criteria:

* Student is 17-20 years of age
* Student is an LMU incoming first-year college student
* Student has access to a cellular device capable of receiving text messages
* Student's parent or legal guardian has an email address on file at LMU
* Student's parent or legal guardian has a cellular device capable of receiving text messages
* Student's parent or legal guardian received an invitation from the research team to participate
* Student's parent or legal guardian signed up to access the assigned intervention
* Student's parent or legal guardian is a resident of the United States
* Informed consent (or assent, as applicable) is provided

Exclusion Criteria:

* Student is not 17-20 years of age
* Student is not an LMU incoming first-year college student
* Student does not have access to a cellular device capable of receiving text messages
* Student's parent or legal guardian does not have an email address on file at LMU
* Student's parent or legal guardian does not have a cellular device capable of receiving text messages
* Student's parent or legal guardian did not receive an invitation from the research team to participate
* Student's parent or legal guardian did not sign up to access the assigned intervention
* Student's parent or legal guardian is not a resident of the United States
* Informed consent (or assent, as applicable) is not provided

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Drinking between Baseline and 3 Months | baseline, 3 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change in Daily Drinking between Baseline and 6 Months | baseline, 6 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change in Peak Drinking Occasion between Baseline and 3 Months | baseline, 3 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change in Peak Drinking Occasion between Baseline and 6 Months | baseline, 6 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change in Heavy Episodic Drinking Occasion between Baseline and 3 Months | baseline, 3 months
  Self-reported number of times 4/5 drinks (female/male) were consumed in a 2-hour period in the past 30 days.
Change in Heavy Episodic Drinking Occasion between Baseline and 6 Months | baseline, 6 months
  Self-reported number of times 4/5 drinks (female/male) were consumed in a 2-hour period in the past 30 days.
Change in Frequency of Intoxication Events between Baseline and 3 Months | baseline, 3 months
  Self-reported number of times individuals reported drinking to intoxication in the past 30 days.
Change in Frequency of Intoxication Events between Baseline and 6 Months | baseline, 6 months
  Self-reported number of times individuals reported drinking to intoxication in the past 30 days.
Change in Number of Alcohol-Related Consequences between Baseline and 3 Month | baseline, 3 months
  Self-reported number of alcohol-related consequences in the past 30 days.
Change in Number of Alcohol-Related Consequences between Baseline and 6 Month | baseline, 6 months
  Self-reported number of alcohol-related consequences in the past 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Marymount, Los Angeles, California, United States